CLINICAL TRIAL: NCT03323957
Title: Development and Evaluation of a New Infant Nutrition Screening Tool
Acronym: iNEWS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Glasgow (Other)
Collaborators: National Health Service, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Dr Konstantinos Gerasimidis, Senior Lecturer in Clinical Nutrition, University of Glasgow
Other Study IDs: 10/S0709/45
Record Dates: First submitted 2017-10-18; First posted 2017-10-27 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Malnutrition; Paediatric Failure to Thrive
MeSH Terms: conditions — Malnutrition; Failure to Thrive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: all infants admitted for care
  Interventions: Diagnostic Test: nutritional screening tool

INTERVENTIONS:
Diagnostic Test: nutritional screening tool — screening of disease associated malnutrition in sick infants

SUMMARY:
A large number of children experience undernutrition related to or resulting from their illness. The NHS has recently published standards which state that all patients should be screened for undernutrition on admission and periodically during their stay at hospital. Although, recent studies have attempted to develop appropriate nutritional screening tool for children on admission, there is no agreement concerning the most appropriate criteria to be used and they have not been validated for use in infants. The project team have developed a preliminary tool that would be both simple and quick to use in order to identify infants who are either undernourished or at risk of undernutrition on admission and who would benefit from referral for full nutritional assessment by a dietician.

The purpose of this study is establish whether an infant Paediatric Yorkhill Malnutrition Score for infants would be able to distinguish infants who are well-nourished from those undernourished or at risk of undernutrition. The researchers will recruit all newly admitted patients ( 210 infants with low, medium, and high risk of undernutrition) from selected wards at the Royal Hospital for Sick Children Glasgow. The result from the infant screening tool will be compared with the rating using the longer Subjective Global Nutritional Assessment to test the ability of Infant Screening Tool to identify infants at high risk of malnutrition. The researcher will also measure the fat store using skinfolds and will compare the results among those rated high or low risk by the new tool. Finally, the utility of iPYMS score, growth trajectory, body mass index and behaviour questionnaire as predictors of low adiposity and stunting will be compared.

DETAILED DESCRIPTION:
Subjects Participant of the study will be all patients newly admitted to selected wards at the Royal Hospital for Sick Children (and possibly RAH Paisley). An average of 8 patients per day are admitted to the relevant wards and this study will aim to recruit a total of 200 over a 4 month period, after an initial pilot with up to 20 patients.

Recruitment The researcher will identify those patients eligible for screening by visiting the wards. The researcher will give an information leaflet to the patient's carer to introduce and explain the study. The researcher will allow plenty at least an hour for them to consider the study. The researcher will then approach the family and answer any questions. If the carer is happy to participate, the researcher will ask him/her to complete a consent form. A copy of the consent form will be given to the carers and another will be placed in the child's medical notes. The researcher will first complete the iPYMS scoring sheet for each child Discriminant validity will then be tested using body composition measurement using triceps (TSF) and subscapular skinfold thickness and the mid upper arm circumference (MUAC) and SGNA (Subjective Global Nutritional Assessment). To test the concurrent validity, the results from the infant screening tool will be compared with the results of STRONG kids (Screening Tool Risk on Nutritional Status and Grow).

Global Nutritional Assessment for infants (SGNA) The researcher will ask the main carers of patients to complete the eating behavior questionnaire about the infant's diet (type of milk. supplementary feeding and weaning diet), weight loss (poor weight gain), gastrointestinal symptoms,and daily activity. A rough visual assessment of the child's muscle stores and fat will be carried out by the researcher. This is a global nutritional assessment procedure recently validated in paediatric patients (Secker & Jeejeebhoy, 2007). The researcher will extract equivalent items for SGNA about the child's food intake, diarrhoea, vomiting, weight loss or poor weight gain or no weight gain, during the few days before admission. An observational assessment of patients will be also carried out by the researcher in terms of diminished subcutaneous fat, muscle mass and hollow face (subjective clinical assessment the same as d). In addition, the researcher will use information recorded in the medical notes of the patient to assess patients' underlying illness with a risk of malnutrition (Anorexia nervosa, Celiac disease, Cystic fibrosis, cardiac disease, and trauma).

Infant EBQ This questionnaire has been developed using population data from a cohort study and is designed to identify infants at risk of weight faltering. This will be completed by the main carers of patients to assess the patient's general appetite and eating behaviour.

Bioelectrical impedance (BIA) This has been developed for assessment of nutritional status in children based on indices of lean and fat adjusted for body size. This study will explore whether this method is practical and effective in this young age range and how it relates to nutrition score.

Length of hospital stay as a secondary outcome will also be collected from hospital admissions statistics or through the notes. Patients' birth weight will be collected by the maternal report in order to calculate weight trajectory

Power Calculation 70 subjects in each group gives 80% power to detect a difference of 0.5 SD in any of the measures between any two of the groups. This study thus aim to recruit 210-250 subjects.

Analysis The data will be used to test the utility of PYMS score, growth trajectory, body mass index and behaviour questionnaire as predictors of low adiposity and stunting.

ELIGIBILITY:
Inclusion Criteria:

- All infant patients admitted to hospital overnight or longer on medical and general surgical wards

Exclusion Criteria:

* Patients in the short stay ward, intensive care or high dependency unit, oncology unit, critical care and cardiology
* Patients who have been transferred from neonatal units and critical care

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participant of the study will be all patients newly admitted to selected wards (medical and general surgical wards) at the Royal Hospital for Sick Children. An average of 8 patients per day are admitted to the relevant wards and we will aim to recruit a total of 250. Children aged 1 -12 months are the subjects of this study as the purpose of this study is to develop a screening tool for infants.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2010-10-01 (Actual); Primary Completion 2017-11-30 (Estimated); Study Completion 2017-11-30 (Estimated)

PRIMARY OUTCOMES:
Mean skinfold z-score | baseline
  The average of triceps (TSF) and subscapular skinfold thickness z-scores (SD) will be calculated as a measure of current nutritional status

SECONDARY OUTCOMES:
Hospital Stay | The period in days from the date of hospital admission until the date of hospital discharge, assessed up to 100 days
  Length of Hospital Stay
Global Nutritional Assessment | baseline
  Global Nutritional Assessment for infants (Subjective Global Nutritional Assessment) as a measure of current and future nutrition risk (well-nourished, moderately malnourished, or severely malnourished).

CONTACTS AND LOCATIONS:
Locations (1):
- New Lister Building, Glasgow Royal Infirmary, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
not allowed from the IPR approval to share data with third parties

REFERENCES:
- [Derived] Gerasimidis K, Milani S, Tester A, Purcell O, Woodley C, Tsiountsioura M, Koulieri A, Zerva O, Loizou K, Rafeey M, Kontogianni M, Wright C. A multicentre development and evaluation of a dietetic referral score for nutritional risk in sick infants. Clin Nutr. 2019 Aug;38(4):1636-1642. doi: 10.1016/j.clnu.2018.08.017. Epub 2018 Sep 5. PMID 30224303

DOCUMENTS (1):
  • Study Protocol (2010-09-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT03323957/Prot_000.pdf